CLINICAL TRIAL: NCT04295499
Title: Clinical Performance of Qualis Silicone Hydrogel Soft Contact Lens Over 3 Months of Daily Wear
Brief Title: Safety and Effectiveness of the Qualis Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unicon Optical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US-PRO1904001
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Device: Qualis Silicone Hydrogel Soft Contact Lens (Experimental): Test lenses will be worn on a daily wear basis for up to one month with removal for cleaning, disinfection, and storage prior to sleeping. Subjects will be instructed to wear the test lenses at least 6 hours a day, a minimum of 5 days per week. The Test Device is investigational and not cleared/approved by the US FDA.
  Interventions: Device: soft (hydrophilic) contact lens
- Control Device: Acuvue Vita Monthly Contact Lens (Active Comparator): Test lenses will be worn on a daily wear basis for up to one month with removal for cleaning, disinfection, and storage prior to sleeping. Subjects will be instructed to wear the test lenses at least 6 hours a day, a minimum of 5 days per week. The Control Device is cleared by the US FDA.
  Interventions: Device: soft (hydrophilic) contact lens

INTERVENTIONS:
Device: soft (hydrophilic) contact lens — The intervention is a daily wear soft contact lens

SUMMARY:
Three-month, open-label, bilateral, parallel group, randomized, daily wear contact lens dispensing study.

DETAILED DESCRIPTION:
Three-month, open-label, bilateral, parallel group, randomized, daily wear contact lens dispensing study comparing the Qualis Silicone Hydrogel Soft Contact Lens for Daily Wear with the currently marketed Acuvue Vita (senofilcon C) Monthly Contact Lens (FDA cleared under K160212). Eligible subjects will be examined for baseline evaluation and lens fitting. Up to fifty (50) subjects will wear the test contact lenses and up to twenty-five (25) subjects will wear the control contact lenses. The subjects will undergo standard ophthalmic evaluation for contact lens wear and will be followed for a period of at least ninety (91) days.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the informed consent form and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 years of age.
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 in each eye.
* The subject's refractive cylinder must be ≤ 0.75 Diopters in each eye.
* The subject must have best corrected visual acuity of 20/25 (LogMAR) or better in each eye.
* Subjects should own a wearable pair of spectacles.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week

Exclusion Criteria:

Subjects may not be enrolled into the study if ANY of the following apply:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
* The use of systemic or ocular medications that would contraindicate contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser in situ keratomileusis (LASIK), etc.).
* Any grade 2 or greater slit lamp findings for corneal staining, and any grade 3 or greater slit lamp findings for other abnormalities (e.g., edema, corneal neovascularization, tarsal abnormalities, conjunctival injection) on the ISO 11980 classification scale, any current inflammatory events or events within the last 6 months, or any other ocular abnormality that may contraindicate contact lens wear.
* Any known hypersensitivity or allergic reaction to Biotrue or ClearCare contact lens care solutions
* Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Extended wear, monovision or multi-focal contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
* Any subject where the randomized lens demonstrates a fit that is deemed inappropriate by the investigator, including, but not limited to, the lens being too flat, too steep, have excessive or inadequate movement, and/or insufficient limbal coverage.
* Employee or relative of employees of sponsor or investigational clinic (e.g., Investigator, Coordinator, Technician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ala Moana Advanced Eye Clinic, Honolulu, Hawaii
  - SUNY College of Optometry, New York, New York
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period started in July 2020 and was closed in October 2020 after successfully fulfilling the enrollment goal (75 subjects). Data collection occurred from July 22, 2020 to January 28, 2021.
Period: Overall Study
Arm/Group | Test Device: Qualis Silicone Hydrogel Soft Contact Lens | Control Device: Acuvue Vita Monthly Contact Lens
Started | 50 (July 22, 2020) | 25 (July 22, 2020)
Completed | 48 (January 28, 2021) | 25 (January 28, 2021)
Not Completed | 2 | 0
Not completed — moving out of state | 1 | 0
Not completed — traveling overseas for business prior to the study completion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Device: Qualis Silicone Hydrogel Soft Contact Lens | Control Device: Acuvue Vita Monthly Contact Lens | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Mean (Full Range); unit: years] | 26.90 [18 to 44] | 27.32 [20 to 43] | 27.04 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 17 | 50
  Male | 17 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 20 | 10 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 14 | 41
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Non-Serious Adverse Reactions
Description: The primary safety endpoint in this evaluation is the rate of serious adverse reactions related to visual acuity loss as well as accompanying slit-lamp findings and other associated observations.
Time Frame: 91 days
Population: open-label, multi-center, randomized concurrent-control study with the treatment duration of 91 days.
  Seventy-five (75) subjects were enrolled in the study-of which 50 subjects wore the test lenses (Qualis (Linofilcon A) Silicone Hydrogel Soft Contact Lens for Daily Wear) and 25 subjects wore the control lenses (Acuvue Vita (senofilcon C) Monthly Contact Lens).
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Test Device: Qualis Silicone Hydrogel Soft Contact Lens | Control Device: Acuvue Vita Monthly Contact Lens
Number analyzed (Participants) | 50 | 25
Number analyzed (eyes) | 100 | 50
eyes
  Non-ocular adverse events (significant but non-serious) | 1 | 3
  Non-device related ocular adverse events (significant but non-serious) | 7 | 0
  Device related ocular adverse events (significant but non-serious) | 1 | 1

2. Primary Outcome: Number of Eyes With Best-corrected Contact Lens Visual Acuity of +0.10 logMAR or Better
Description: The primary efficacy endpoint in this evaluation is the percentage of subjects with best-corrected contact lens visual acuity of +0.10 logMAR or better
Time Frame: 91 days
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Test Device: Qualis Silicone Hydrogel Soft Contact Lens | Control Device: Acuvue Vita Monthly Contact Lens
Number analyzed (Participants) | 50 | 25
Number analyzed (eyes) | 100 | 50
eyes
  Initial best corrected contact lens visual acuity with spherical over-refraction | 100 | 50
  Visual acuity (VA) results -Day91- | 96 | 47

ADVERSE EVENTS:
Time Frame: through study completion, every visit, Day7,Day 14,Day 30, Day 60 and Day 91.
Description: Through study completion, every visit, Day7,Day 14,Day 30, Day 60 and Day 91. by regular investigator assessment. In general, an 'adverse event' refers to any undesirable clinical occurrence in a subject, whether it is considered to be device-related or not.
Arm/Group | Test Device: Qualis Silicone Hydrogel Soft Contact Lens | Control Device: Acuvue Vita Monthly Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 6/50 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Device: Qualis Silicone Hydrogel Soft Contact Lens (N=50) | Control Device: Acuvue Vita Monthly Contact Lens (N=25)
Common cold (General disorders) | 0 (0) | 1 (1) — Common cold - not COVID-19; confirmed by PCR testing.
Migraines (General disorders) | 1 (1) | 0 (0) — Migraines
Covid-19 positive (General disorders) | 0 (0) | 2 (2) — Covid-19 positive.
Presceptal Cellulitis (Eye disorders) | 1 (1) | 0 (0) — Presceptal Cellulitis, right eye
Internal hordeolum (Eye disorders) | 1 (1) | 0 (0) — Internal hordeolum, right eye
Visual aura (Eye disorders) | 1 (1) | 0 (0) — Visual aura associated with migraine headaches. OU
papillary conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — papillary conjunctivitis, right eye
Mild contact dermatitis (Eye disorders) | 1 (1) | 0 (0) — Mild contact dermatitis, OU

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04295499/Prot_SAP_003.pdf
  • Informed Consent Form (2020-06-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT04295499/ICF_002.pdf